CLINICAL TRIAL: NCT00758160
Title: From Immediate-release MPH to OROS MPH: The Impact Upon Family of Children and Adolescents With ADHD
Brief Title: The Impact of Osmotic Release Oral Delivery System Methylphenidate (OROS MPH) Upon Family of Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015331; CONCERTAATT4086; CCT-TWN-MA6
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder With Hyperactivity; Methylphenidate; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OROS methylphenidate (Experimental): Participants willl receive Osmotic Release Oral Delivery System (OROS) methylphenidate (MPH) 18 milligram (mg), 36 mg or 54 mg once daily for 8 weeks. Dose will be adjusted for each participant based on clinical responses and/or side effects.
  Interventions: Drug: OROS Methylphenidate

INTERVENTIONS:
Drug: OROS Methylphenidate — Participants will receive Osmotic Release Oral Delivery System (OROS) methylphenidate (MPH) 18 milligram (mg), 36 mg or 54 mg once daily for 8 weeks. Dose will be adjusted for each participant based on clinical responses and/or side effects.

SUMMARY:
The purpose of this study is to evaluate whether familial relationships and psychological status of participants or caregivers as well as Attention Deficit Hyperactivity Disorder (ADHD) symptoms of participants can be improved by switching from Immediate-release Methylphenidate (IR-MPH) to Osmotic Release Oral Delivery System Methylphenidate (OROS-MPH).

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), single-arm, open-label (all people know the identity of the intervention), 8-week, multi-centric (conducted in more than 1 center) study. OROS-MPH will be administered orally for 2 months at doses of 18, 36, or 54 milligram (mg) to replace IR-MPH. Clinicians will adjust the dose of each participant according to participant's clinical responses and/or side effects. During the study period, participants will be assessed on Week 2, 4, and 8. Efficacy will be evaluated primarily based on change from baseline in Chinese version of the 26-item Swanson, Nolan and Pelham-Fourth Edition (SNAP-IV) rating scale assessed by parents and Chinese Health Questionnaire (CHQ). Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Participants who have been treated with Immediate-release methyphenidate (IR-MPH) for at least 4 weeks before enrollment, but previous treatment is considered unsatisfactory due to 1 or more of the following reasons: lack of effectiveness, lack of tolerability or safety, lack of compliance, and/or other reasons
* Participants who are able to comply with the study visit schedule and whose parents/caregiver and community school teacher are willing and able to complete the protocol-specified assessments
* Participants who are still at school
* Participants who are treated with greater than equal to 10 milligram (mg) IR-MPH daily before enrollment

Exclusion Criteria:

* Participants who cannot understand or follow the instructions given in the study
* Participants with serious or unstable medical illness
* Participants who have clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract
* Participants who have glaucoma (increased pressure inside the eye that causes visual problems), an ongoing seizure disorders, or a psychotic disorder
* Participants who are hypersensitive to methylphenidate
* Participants who have any co-existing medical condition or are taking a concomitant medication that is likely to interfere with safe administration of methylphenidate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS MPH: Participants received Osmotic Release Oral Delivery System (OROS) methylphenidate (MPH) 18 milligram (mg), 36 mg or 54 mg once daily for 8 weeks. Dose was adjusted for each participant based on clinical responses and/or side effects.
Period: Overall Study
Arm/Group | OROS MPH
Started | 296
Completed | 230
Not Completed | 66
Not completed — No Longer Requires Study Medication | 4
Not completed — Administration Problems | 3
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 10
Not completed — Lost to Follow-up | 14
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | OROS MPH
Number analyzed (Participants) | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 247

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Swanson, Nolan and Pelham-Fourth Edition (SNAP-IV) Rating Scale (Parents) Score at Week 2
Description: Parents were asked to assess their children on a 26-item Chinese SNAP-IV questionnaire consisting of inattention (items 1-9; subscore range 0-27), hyperactivity (items 10-18; subscore range 0-27) and oppositional (19-26, subscore range 0-24) subscales used to assess the qualitative judgments in Attention Deficit Hyperactivity Disorder (ADHD). Each item was based on a 4-point likert scale ranging from 0 (not at all) to 3 (very much). The overall score ranged from 0 to 78. The total score for Inattention and hyperactivity ranged from 0 to 27 and for oppositional ranged from 0 to 21. Mean Change was calculated as mean SNAP-IV score at Week 2 minus mean SNAP-IV score at Baseline.
Time Frame: Baseline and Week 2
Population: Intent-to-treat (ITT) analysis set included all participants who received OROS-MPH at least once and provided at least 1 post-baseline efficacy measurement. Here, 'n' included those participants who were evaluable for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 296
Units on a scale
  Baseline: Inattention (n = 293) | 1.7 (0.6)
  Baseline: Hyperactivity (n = 293) | 1.4 (0.7)
  Baseline: Oppositional (n = 296) | 1.3 (0.7)
  Change at Week 2: Inattention (n = 293) | -0.4 (0.5)
  Change at Week 2: Hyperactivity (n = 293) | -0.3 (0.5)
  Change at Week 2: Oppositional (n = 296) | -0.3 (0.5)

2. Primary Outcome: Mean Change From Baseline in Swanson, Nolan and Pelham-Fourth Edition (SNAP-IV) Rating Scale (Parents) Score at Week 4
Description: Parents were asked to assess their children on a 26-item Chinese SNAP-IV questionnaire consisting of inattention (items 1-9; subscore range 0-27), hyperactivity (items 10-18; subscore range 0-27) and oppositional (19-26, subscore range 0-24) subscales used to assess the qualitative judgments in Attention Deficit Hyperactivity Disorder (ADHD). Each item was based on a 4-point likert scale ranging from 0 (not at all) to 3 (very much). The overall score ranged from 0 to 78. The total score for Inattention and hyperactivity ranged from 0 to 27 and for oppositional ranged from 0 to 21. Mean Change was calculated as mean SNAP-IV score at Week 4 minus mean SNAP-IV score at Baseline.
Time Frame: Baseline and Week 4
Population: ITT analysis set included all participants who received OROS-MPH at least once and provided at least 1 post-baseline efficacy measurement. Here, 'n' included those participants who were evaluable for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- OROS MPH: Participants received OROS MPH 18 mg, 36 mg or 54 mg once daily for 8 weeks. Dose was adjusted for each participant based on clinical responses and/or side effects.
Arm/Group | OROS MPH
Number analyzed (Participants) | 296
Units on a scale
  Change at Week 4: Inattention (n = 293) | -0.4 (0.6)
  Change at Week 4: Hyperactivity (n = 293) | -0.3 (0.6)
  Change at Week 4: Oppositional (n = 296) | -0.3 (0.6)

3. Primary Outcome: Mean Change From Baseline in Swanson, Nolan and Pelham-Fourth Edition (SNAP-IV) Rating Scale (Parents) Score at Week 8
Description: Parents were asked to assess their children on a 26-item Chinese SNAP-IV questionnaire consisting of inattention (items 1-9; subscore range 0-27), hyperactivity (items 10-18; subscore range 0-27) and oppositional (19-26, subscore range 0-24) subscales used to assess the qualitative judgments in Attention Deficit Hyperactivity Disorder (ADHD). Each item was based on a 4-point likert scale ranging from 0 (not at all) to 3 (very much). The overall score ranged from 0 to 78. The total score for Inattention and hyperactivity ranged from 0 to 27 and for oppositional ranged from 0 to 21. Mean Change was calculated as mean SNAP-IV score at Week 8 minus mean SNAP-IV score at Baseline.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 296
Units on a scale
  Change at Week 8: Inattention (n = 293) | -0.5 (0.6)
  Change at Week 8: Hyperactivity (n = 293) | -0.4 (0.6)
  Change at Week 8: Oppositional (n = 296) | -0.4 (0.6)

4. Primary Outcome: Mean Change From Baseline in Chinese Health Questionnaire (CHQ) at Week 4
Description: The CHQ is a self administered screening instrument used to assess psychiatric morbidity in the Chinese community. It was derived from the General Health Questionnaire, and has been validated with satisfactory construct validity and applied in the survey of psychiatric morbidity in the community and in hospital settings. Four factors are included in the structure: somatic symptoms; anxiety and worrying; sleep problems; and depression and poor family relationships. It contains 12 items, with a maximum score of 12. CHQ scores indicated the severity of participants' psychological problems (0-2=normal; 3-4=minor; 5-6=moderate; and 7-12=severe psychological problems). Mean Change was calculated as mean CHQ score at Week 4 minus mean CHQ score at Baseline.
Time Frame: Baseline and Week 4
Population: ITT analysis set included parents of all the participants who received OROS-MPH at least once and provided at least 1 post-baseline efficacy measurement. 'N' (number of participants analyzed) included those participants who were evaluable for this measure. 'n' included those participants who were evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 275
Units on a scale
  Baseline: Mother Assessment (n = 275) | 1.9 (0.6)
  Baseline: Father Assessment (n = 216) | 1.7 (0.4)
  Change at Week 4: Mother Assessment (n = 275) | -0.1 (0.4)
  Change at Week 4: Father Assessment (n = 216) | 0 (0.3)

5. Primary Outcome: Mean Change From Baseline in Chinese Health Questionnaire (CHQ) at Week 8
Description: The CHQ is a self administered screening instrument used to assess psychiatric morbidity in the Chinese community. It was derived from the General Health Questionnaire, and has been validated with satisfactory construct validity and applied in the survey of psychiatric morbidity in the community and in hospital settings. Four factors are included in the structure: somatic symptoms; anxiety and worrying; sleep problems; and depression and poor family relationships. It contains 12 items, with a maximum score of 12. CHQ scores indicated the severity of participants' psychological problems (0-2=normal; 3-4=minor; 5-6=moderate; and 7-12=severe psychological problems). Mean Change was calculated as mean CHQ score at Week 8 minus mean CHQ score at Baseline.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 275
Units on a scale
  Change at Week 8: Mother Assessment (n = 275) | -0.1 (0.4)
  Change at Week 8: Father Assessment (n = 216) | 0 (0.4)

6. Secondary Outcome: Chinese Version of the Family Adaptation, Partnership, Growth, Affection, and Resolve (Family APGAR-C) Score
Description: Parents of the participants were asked to assess the Family APGAR which is a 5-item questionnaire designed to assess the 5 dimensions of perceived family support: Adaptation, Partnership, Growth, Affection, and Resolve. Each item is rated on a 3-point scale ranging from 0 to 2 where 0=hardly ever, 1=some of the time and 2=almost always. The total score ranges from 0 to 10 with greater scores indicating greater family support.
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 281
Units on a scale
  Baseline: Mother Assessment (n = 275) | 6.4 (2.9)
  Baseline: Father Assessment (n = 216) | 6.5 (2.5)
  Week 4: Mother Assessment (n = 280) | 6.6 (2.8)
  Week 4: Father Assessment (n = 223) | 6.7 (2.5)
  Week 8: Mother Assessment (n = 281) | 6.5 (3)
  Week 8: Father Assessment (n = 226) | 6.6 (2.7)

7. Secondary Outcome: Swanson, Nolan and Pelham-Fourth Edition (SNAP-IV) Rating Scale (Teachers) Score
Description: Teachers were asked to assess the children on a 26-item Chinese SNAP-IV questionnaire consisting of inattention (items 1-9; subscore range 0-27), hyperactivity (items 10-18; subscore range 0-27) and oppositional (19-26, subscore range 0-24) subscales used to assess the qualitative judgments in Attention Deficit Hyperactivity Disorder (ADHD). Each item was based on a 4-point likert scale ranging from 0 (not at all) to 3 (very much). The overall score ranged from 0 to 78. The total score for Inattention and hyperactivity ranged from 0 to 27 and for oppositional ranged from 0 to 21.
Time Frame: Baseline, Week 2, 4 and 8
Population: ITT analysis set included of all the participants who received OROS-MPH at least once and provided at least 1 post-baseline efficacy measurement. 'N' (number of participants analyzed) included those participants who were evaluable for this measure. 'n' included those participants who were evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 288
Units on a scale
  Baseline: Inattention (n = 281) | 1.5 (0.7)
  Baseline:Hyperactivity (n = 285) | 1.1 (0.7)
  Baseline: Oppositional (n = 283) | 0.9 (0.7)
  Week 2: Inattention (n = 286) | 1.3 (0.7)
  Week 2: Hyperactivity (n = 287) | 0.9 (0.7)
  Week 2: Oppositional (n = 286) | 0.7 (0.7)
  Week 4: Inattention (n = 287) | 1.2 (0.6)
  Week 4: Hyperactivity (n = 288) | 0.9 (0.8)
  Week 4: Oppositional (n = 287) | 0.7 (0.7)
  Week 8: Inattention (n = 287) | 1.1 (0.6)
  Week 8: Hyperactivity (n = 288) | 0.8 (0.7)
  Week 8: Oppositional (n = 287) | 0.7 (0.7)

8. Secondary Outcome: Social Adjustment Scale Score for Children and Adolescents (SAICA)
Description: SAICA is a 77-item semi-structured interview scale designed for administration to school-aged children with age 6-18 years, or to their parents about their children. SAICA provides an evaluation of children's current functioning in the domains of school, spare time, peer relations, and home behaviors. Each item ranged on a 4-point likert scale ranging from 1 to 4 with a higher mean score indicating either poorer social function or a more severe social problem.
Time Frame: Baseline, Week 4 and Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 165
Units on a scale
  Baseline (n = 151) | 1.5 (0.7)
  Week 4 (n = 160) | 1.8 (0.3)
  Week 8 (n = 165) | 1.8 (0.3)

9. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Score
Description: CGI-ADHD-S is a single item assessment of the global severity of ADHD symptoms in relation to the clinician's total experience after reviewing all the returned questionnaires and clinical assessment of participants' behavioral symptoms. Severity is rated on a 7-point scale ranging from 1 to 7 with 1=normal (not at all ill) and 7=most extremely ill.
Time Frame: Baseline, Week 2, 4 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 292
Units on a scale
  Baseline (n = 290) | 4.3 (0.9)
  Week 2 (n = 291) | 3.5 (1.0)
  Week 4 (n = 291) | 3.1 (1.1)
  Week 8 (n = 292) | 3.0 (1.1)

10. Secondary Outcome: Number of Participants With Clinical Global Impression-Improvement (CGI-I) Score
Description: CGI-I is a single item assessment of the global improvement of ADHD symptoms in relation to the clinician's total experience after reviewing all the returned questionnaires and clinical assessment of participants' behavioral symptoms. Improvement is rated on a 7-point scale (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse).
Time Frame: Baseline, Week 2, 4 and 8
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | OROS MPH
Number analyzed (Participants) | 292
Participants
  Week 2: Very much improved (n = 292) | 4
  Week 2: Much improved (n = 292) | 98
  Week 2: Minimally improved (n = 292) | 126
  Week 2: No change (n = 292) | 45
  Week 2: Minimally worse (n = 292) | 16
  Week 2: Much worse (n = 292) | 2
  Week 2: Very much worse (n = 292) | 1
  Week 4: Very much improved (n = 262) | 15
  Week 4: Much improved (n = 262) | 111
  Week 4: Minimally improved (n = 262) | 96
  Week 4: No change (n = 262) | 27
  Week 4: Minimally worse (n = 262) | 10
  Week 4: Much worse (n = 262) | 3
  Week 4: Very much worse (n = 262) | 0
  Week 8: Very much improved (n = 282) | 16
  Week 8: Much improved (n = 282) | 129
  Week 8: Minimally improved (n = 282) | 91
  Week 8: No change (n = 282) | 28
  Week 8: Minimally worse (n = 282) | 13
  Week 8: Much worse (n = 282) | 4
  Week 8: Very much worse (n = 282) | 1

11. Secondary Outcome: Global Assessment of Satisfaction by Parents/Caregivers
Description: Parents/caregivers were asked to assess the satisfaction with respect to ADHD treatment on a 5-point scale ranging from 1 to 5 where 1=completely dissatisfied, 2=somewhat dissatisfied, 3=neutral, 4=somewhat satisfied, and 5=completely satisfied.
Time Frame: Baseline, Week 2, 4 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 291
Units on a scale
  Baseline (n = 290) | 3.1 (0.9)
  Week 2 (n = 291) | 3.4 (0.8)
  Week 4 (n = 291) | 3.7 (0.8)
  Week 8 (n = 291) | 3.6 (0.9)

12. Other Pre Specified Outcome: Global Assessment of Satisfaction by Participant
Description: Participants were asked to assess their satisfaction with respect to ADHD treatment on a 5-point scale ranging from 1 to 5 where 1=completely dissatisfied, 2=somewhat dissatisfied, 3=neutral, 4=somewhat satisfied and 5=completely satisfied.
Time Frame: Baseline, Week 2, 4 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS MPH
Number analyzed (Participants) | 291
Units on a scale
  Baseline (n = 290) | 3.2 (0.9)
  Week 2 (n = 291) | 3.5 (0.8)
  Week 4 (n = 291) | 3.7 (0.8)
  Week 8 (n = 291) | 3.6 (0.9)

ADVERSE EVENTS:
Description: Adverse events(AEs) data was reported for each visit as total data for AEs were not analyzed. In addition to the AEs reported in the below table, a category of AEs titled "Other" was reported as no dictionary was used and events under this category were not further specified. Total # affected by other AEs is minimum number of participants affected.
Groups:
- OROS MPH-Baseline; OROS MPH-Week 2; OROS MPH-Week 4; OROS MPH-Week 8: Participants received Osmotic Release Oral Delivery System (OROS) methylphenidate (MPH) 18 milligram (mg), 36 mg or 54 mg once daily for 8 weeks. Dose was adjusted for each participant based on clinical responses and/or side effects.
Arm/Group | OROS MPH-Baseline | OROS MPH-Week 2 | OROS MPH-Week 4 | OROS MPH-Week 8
Serious Adverse Events (participants affected / at risk) | 0/296 | 0/296 | 0/296 | 0/296
Other Adverse Events (participants affected / at risk) | 80/296 | 100/296 | 90/296 | 95/296
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS MPH-Baseline (N=296) | OROS MPH-Week 2 (N=296) | OROS MPH-Week 4 (N=296) | OROS MPH-Week 8 (N=296)
Appetite decreased (General disorders) | 80 | 100 | 90 | 95
Nausea (General disorders) | 22 | 22 | 15 | 15
Insomnia (General disorders) | 22 | 35 | 30 | 25
Headache (General disorders) | 17 | 14 | 8 | 7
Dizziness (General disorders) | 12 | 10 | 6 | 9
Somnolence (General disorders) | 8 | 4 | 2 | 1
Abdominal pain (General disorders) | 17 | 20 | 11 | 12
Stomachache (General disorders) | 5 | 4 | 1 | 1
Other (General disorders) | 26 | 32 | 25 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less